CLINICAL TRIAL: NCT00571194
Title: A Single-dose Pilot Study to Evaluate the Pharmacokinetics of Pravastatin Given as an Oral Dose in Pediatric and Adolescent Subjects 12 Months to 16 Years of Age Receiving Continuous Cycling Peritoneal Dialysis
Brief Title: Single Dose Pravastatin Pharmacokinetics in Pediatric Peritoneal Dialysis Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 75611
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: End Stage Renal Disease
Keywords: pravastatin, peritoneal dialysis, pediatric patients
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Pravastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- peritoneal dialysis (CCPD) (Other): PK profile of pravastatin
  Interventions: Drug: pravastatin

INTERVENTIONS:
Drug: pravastatin — A single 10 mg dose of pravastatin will be administered 3 mL blood samples for pravastatin Pharmacokinetic evaluations will be collected at 0.5, 1, 2, 3, 4, 6, and 8 hours. 5 mL blood samples for pravastatin PK and laboratory evaluations will be drawn at pre-dose and 24 hours.
  Vital Signs and Physical Exams will also be done throughout the study
  Other Names: Pravachol

SUMMARY:
Many children with end stage renal disease develop hyperlipidemia. HMG-CoA (3-hydroxy-3-methylglutaryl-coenzyme A) reductase inhibitors, such as pravastatin, are typical treatments for hyperlipidemia. However, we do not know how pravastatin is metabolized in patients on dialysis. This study is designed to provide preliminary pharmacokinetic data for pravastatin in pediatric patients on peritoneal dialysis.

DETAILED DESCRIPTION:
This is a single-dose pilot study to evaluate the pharmacokinetic profile of pravastatin in 7 pediatric and adolescent subjects ranging from 12 months to 16 years of age who are on dialysis. The study group will be comprised of healthy children receiving continuous cycling peritoneal dialysis (CCPD). Pravastatin dosing will be 10 mg in all subjects. Blood, urine, and dialysate samples will be obtained over a 24-hour period post-dose for measurement of pravastatin concentrations. Safety evaluations will include adverse events (AEs), physical examination, vital signs, and clinical laboratory evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from 12 months to 18 years of age.
2. Patients with end stage renal disease who receive continuous cycling peritoneal dialysis.
3. signed informed consent
4. Physical exam demonstrates no abnormalities that would make this study medically hazardous to the subject.

   -

Exclusion Criteria:

1. Any clinically significant unstable medical condition or chronic disease other than those associated with ESRD.
2. Any clinically significant illness within 10 days or receiving single-sdoe of study medication
3. History of rhabdomyolysis
4. Clinically significant liver disease or history of malabsorption or previous gastrointestinal surgery that could effect drug absorption or metabolism.
5. Clinical laboratory abnormalities: Aspartate aminotransferase (AST), Alanine Aminotransferase (ALT), Creatine phosphokinase(CPK) > 2.5 times upper limit of normal; hemoglobin < 8.5 g.dL.
6. Known hypersensitivity to pravastatin
7. Unwilling to have blood samples drawn
8. Has taken a HMG-CoA reductase inhibitor in the last week -

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eileen N Ellis, MD, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share the data

RESULTS

PARTICIPANT FLOW:
Groups:
- Pravastatin: Study drug given and have levels done to measure pharmacokinetics.
Period: Overall Study
Arm/Group | Pravastatin
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- A Single-Dose Pilot Study: Study drug given and have levels done to measure pharmacokinetics
Arm/Group | A Single-Dose Pilot Study
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics
Time Frame: 24 hours
Population: Data was not collected
Arm/Group | A Single-Dose Pilot Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | A Single-Dose Pilot Study
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes